CLINICAL TRIAL: NCT05835947
Title: The Role of Early Detection and Treatment of Anal Intraepithelial Neoplasia in the Prevention of Anal Squamous Cell Carcinoma in Women: Establishing the Disease Burden in Women With Genital Cancer
Brief Title: Anal Cancer Risk In Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 315094
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Anal Cancer; Human Papilloma Virus; Anal Intraepithelial Neoplasia; Genital Neoplasm; Genital Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dual Pathology — Women with both genital HSIL/SCC and Anal HSIL/SCC

SUMMARY:
This is a retrospective cross-sectional study involving the analysis of Cancer Registry Data. As part of this study, cancer registration data collated by the National Cancer Registration and Analysis Service (NCRAS; the national cancer registry in England), via NHS Digital data access request service (DARS), will be analysed on all female patients aged between 25-90+ years in England with a registered diagnosis of anal and vaginal and/or vulvar and/or cervical cancer and/or high grade squamous intraepithelial lesions (HSIL) between 2001 and 2019. For these patients information on age at diagnosis, ethnicity, deprivation, performance status, stage of the cancer at diagnosis, the date of each diagnosis, the treatment received for the diagnosis and the route to diagnosis, will be analysed. Additionally, the total number of women/year (between 1995 and 2019), in England, aged between 25-90+ years with a diagnosis of anal, vulvar, vaginal and cervical cancer as well as their respective HSILs will be requested. Together this data will be used to establish the incidence of anal cancer and HSIL in women with genital cancers and/or HSILs, the progression timelines between the different pathologies, as well as identify relevant sociodemographic risk factors in this patient group.

DETAILED DESCRIPTION:
Hypothesis: Women with genital HSILs/SCCs have an increased risk of anal HSIL/SCC regardless of whether they have received treatment for their genital condition and would benefit from surveillance and treatment of anal HSIL in the prevention of ASCC.

This is a retrospective observational (cross sectional) study in which de-personalised patient level National Cancer Registration and Analysis Service data via NHS Digital DARS will be requested.

In particular, patient level data for all women in England, between 2001 and 2019, aged 25- 90+ years, with a diagnosis of anal cancer and/or anal HSIL and:

* vaginal SCC and/or HSIL
* vulvar SCC and/or HSIL
* cervical SCC and/or HSIL
* vaginal and vulvar SCC and/or HSIL
* vaginal and cervical SCC and/or HSIL
* vulvar and cervical SCC and/or HSIL
* vaginal, cervical and vulvar SCC and/or HSIL

For these women with synchronous or metachronous anal and genital HSILs or SCCs data will be collected on:

1. Month, Year of each diagnosis.
2. Age at each diagnosis.
3. Cancer stage (for each cancer): 1, 2, 3, 4, not known, other, unstageable disease.
4. Performance status at each diagnosis: 1,2,3,4, not known.
5. Treatments received (for each diagnosis): Surgery, Chemotherapy, Radiotherapy.
6. Ethnicity: British, Irish, Other white, White/ Black Caribbean, White/Black African, White/ Asian, Other Mixed, Indian, Pakistani, Bangladeshi, Other Asian, Black Caribbean, Black African, Other black, Chinese, Other Ethnic, Not Known.
7. Route to Diagnosis (for each diagnosis): Emergency Presentation, GP referral, Inpatient Elective, Other Outpatient, Screening, Two Week Wait, Unknown.
8. Deprivation score: 1 (least deprived), 2, 3, 4, 5 (Most deprived).

In order to establish the incidence of anal cancer in women with genital cancers, data will be requested on the total number of women/year (between 2001 and 2019), in England, aged between 25-90+ years with a diagnosis of:

* Anal cancer
* Anal HSIL
* Vulvar cancer
* Vulvar HSIL
* Vaginal cancer
* Vaginal HSIL
* Cervical cancer
* Cervical HSIL

ICD-10 malignant neoplasm and carcinoma in-situ codes will be used to identify these patients:

* Anal Cancer C21.0. C21.1, C21.8
* Cancer of the Vulva C51.0, C51.1, C51.2, C51.8, C51.9
* Cancer of the Vagina C52.
* Cancer of the Cervix Uteri C53.0, C53.1, C53.8, C53.9
* Anal HSIL D01.3
* Vulval HSIL D07.1
* Vaginal HSIL D07.2
* Cervical HSIL D06.0, D06.1, D06.7, D06.9

Primary Objective:

Establish the incidence of anal HSIL and cancer in women with genital HSILs and/cancers and vice versa in England.

Secondary Objectives:

1. Asses the risk of anal HSIL and SCC in women with genital HSILs and/or SCC in England.
2. Investigate the sociodemographic risk profile of women developing multizonal anogenital HPV driven high-risk pathologies.
3. Establish the timelines between the development of genital HSIL/SCC and anal HSIL/SCC.

Primary Outcome:

The incidence of anal HSIL and cancer in women with genital HSIL and/cancer in England between 2001- 2019.

Secondary Outcomes:

1. The risk of anal HSIL and/or SCC in women with genital HSILs and/or SCC in England.
2. The relationship between the incidence of multizonal anogenital disease and specific sociodemographic risk factors (ethnicity, age, social deprivation).
3. The amount of time in years and months between the diagnosis of genital HSIL/SCC and anal HSIL/SCC.

Statistics and Data Analysis:

Data will be analysed using SPSS Statistics software. All outcomes extracted from the database will be expressed in categorical fields; therefore, comparisons of outcomes will be analysed using Chi squared or Fisher's Exact Tests. A statistically significant p value for this analysis is defined as p < 0.05. Incidence will be calculated per 100,000 people per year. Any missing data fields were classified as "unknown" within the database. Missing data will not be excluded from the analysis and "unknown" variables are included with tables and figures to prevent bias.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-90+ years of age.
* Women diagnosed with anal cancer and/or HSIL between 2001 and 2019.
* The anogenital cancer must be a squamous cell carcinoma.
* Women with a diagnosis of anal cancer and/or HSIL and:

  1. vaginal cancer and/ or HSIL
  2. vulvar cancer and/or HSIL
  3. cervical cancer and/or HSIL
  4. vaginal and vulvar cancer and/or HSIL
  5. vaginal and cervical cancer and/or HSIL
  6. vulvar and cervical cancer and/or HSIL
  7. vaginal, cervical and vulvar cancer and/or HSIL

Exclusion Criteria:

* Men with a diagnosis of anal HSIL and/or SCC.
* Women aged outside of the 25-90+ years bracket.
* Women diagnosed with anal cancer or HSIL before 2001 and after 2019.
* Women with genital or anal cancer which is not a squamous cell carcinoma.

Ages: 25 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in England affected by both an anal and a genital HSILs/SCCs between 2001-2019.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of anal HSIL and cancer in women with genital HSIL and/cancer in England | 2001- 2019
  as above

SECONDARY OUTCOMES:
he risk of anal HSIL and/or SCC in women with genital HSILs and/or SCC in England | 2001-2019
  as above
The relationship between the incidence of multizonal anogenital disease and specific sociodemographic risk factors. | 2001-2019
  as above
The amount of time in years and months between the diagnosis of genital HSIL/SCC and anal HSIL/SCC | 2001-2019
  as above

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Request to NHS digital is for de-personalised data. Researchers will not have access to individual participant data.